CLINICAL TRIAL: NCT07145840
Title: A Study of Suicidal Behavior Among Schizophrenic Patients
Brief Title: Suicidal Behavior Among Schizophrenic Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, asmaa, Resident of Neuropsychiatry Department, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 35394/4/22
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Suicidal Behavior; Schizophrenic Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients with schizophrenia. They had a current history of suicide ideation or attempt.
  Interventions: Other: Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
- Group B: Patients with schizophrenia without any history of neither suicide ideation nor attempt.
  Interventions: Other: Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)

INTERVENTIONS:
Other: Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) — Psychiatric interview for diagnosis of schizophrenia by SCID 5 (American Psychiatric Association, 2015), The Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) is a semi structured interview guide for making the major DSM-5 diagnoses using the chapter of schizophrenia spectrum

SUMMARY:
This study aimed to; -

1. Study suicidal behavior among sample of schizophrenic patients.
2. Study relation between schizophrenic symptoms and suicidal behavior.
3. Study the relation of mood symptoms in schizophrenic patients and suicidal behavior.

DETAILED DESCRIPTION:
Suicide is a major public health concern. According to the World Health Organization (WHO), approximately one million people die by suicide each year worldwide. This statistic means that every 40 seconds, someone dies by suicide somewhere on the globe, with many more people making non-lethal suicide attempts. It has been suggested that the number of individuals who attempt suicide without causing death is about 10-15 times the number of those who die by suicide.

Schizophrenia is a severe psychiatric disorder characterized by cognitive impairment and behavioral dysfunction. Patients with schizophrenia are at an elevated risk of self-harm, suicide, and all-cause mortality, which results in a reduction of life expectancy of up to 20 years compared with the general population.

Suicide risk in schizophrenia is notably high, and early detection depends on recognizing and evaluating clinical manifestations of depression, despair, and hopelessness, as well as the nature and severity of the psychotic experience, particularly in recently diagnosed patients with higher cognitive function and educational backgrounds.

There is a lack of studies on suicidal behaviors in schizophrenic patients in Arab countries. A study on overall suicidality in Arab countries reported a lifetime suicide attempt rate of 0.72%-6.3% and a suicide ideation rate of 2.09%-13.9%. More research is needed in this area due to the societal and economic costs of suicidal behavior in schizophrenic patients. This issue is a high priority for public health. Several trials have aimed to identify valid predictors of suicide risk. These predictors could not only help reduce the mortality associated with suicidality but also enable a more rational allocation of resources for treatment. Previous suicide attempts, depressive symptoms, hopelessness, and akathisia have been identified as reliable predictors of suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60.
2. Both females and males will be included.
3. All patients should meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for schizophrenia.

Exclusion Criteria:

1. Any neurological disorder.
2. Past history of head trauma.
3. Medical or autoimmune disorders.
4. Other psychiatric disorders e. g. bipolar disorders, post-traumatic stress disorder (PTSD), obsessive compulsive disorder (OCD), and anxiety.
5. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This cross-sectional study was carried out on patients diagnosed with schizophrenia recruited from inpatient and outpatient services of the Department of Neuropsychiatry and Center of Psychiatry, Neurology, Tanta University Hospitals, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Severity of Suicidal Ideation | Within 1 week prior to assessment
  Assessed using the Arabic version of the Beck Scale for Suicide Ideation (BSS), which includes 21 statement groups rated on a 3-point scale. The total score ranges from 0 to 38, with higher scores indicating more severe suicidal ideation.

SECONDARY OUTCOMES:
Severity of Schizophrenia Symptoms | Within 7 days
  Measured using the Positive and Negative Syndrome Scale (PANSS), which assesses positive, negative, and general psychopathology symptoms. Higher scores reflect greater symptom severity.
Severity of Depressive Symptoms | Within 7 days
  Measured using the Arabic version of the Hamilton Depression Rating Scale (HDRS-17). Total scores classify depression as mild, moderate, severe, or very severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.